CLINICAL TRIAL: NCT03775577
Title: Exercise Intolerance in Heart Failure: the Role of Altered Cardiac and Skeletal Muscle Energetics
Brief Title: Exercise Intolerance in Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00129787; R01HL061912 (NIH)
Record Dates: First submitted 2018-11-01; First posted 2018-12-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Heart Failure with Preserved Ejection Fraction; HFpEF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HFpEF: Participants with Heart Failure with Preserved Ejection Fraction
- HFrEF: Participants with Heart Failure with Reduced Ejection Fraction
- Hypertensive Subjects: Participants with Hypertension
- Healthy Subjects: Participants without heart failure and without commodities

SUMMARY:
The investigators are studying whether metabolic abnormalities in cardiac and skeletal muscle in patients with heart failure with preserved ejection fraction (HFpEF) are associated with debilitating exercise intolerance.

DETAILED DESCRIPTION:
This research is being done to better understand why patients with heart failure have difficulty exercising and performing some activities of daily living. Heart muscle and skeletal muscle (in the legs and arms) depend on normal metabolism (the conversion of foods to chemical fuel) to function properly. Investigators will measure metabolites in the heart and leg muscles, including the levels of high energy phosphates and lipids (fats) using magnetic resonance (MR) techniques. High-energy phosphates serve as a source of energy, which is used by the heart and skeletal muscle for contraction. Magnetic resonance uses magnetic fields to measure the levels of these substances.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender who are greater than 21 years of age (no upper age limit),
* Permission of patient's clinical attending physician,
* Previous clinical diagnosis of HF with current New York Heart Association (NYHA) Class II-III symptoms for at least 1 month,
* Left ventricular ejection fraction (EF) >50% by echocardiography, MRI, CT or x-ray or nuclear ventriculography within prior 12 months,
* Stable medical therapy for at least 30 days (no addition or removal or major (>100%) dose change of Renin-Angiotensin-Aldosterone System (RAAS) antagonists, beta-blockers, or calcium channel blockers for hypertension).

Exclusion Criteria:

* Unable to understand the risks, benefits, and alternatives of participation and give meaningful consent,
* Contraindications to MRI such as implanted metallic objects (pre-existing cardiac pacemakers, cerebral clips) or indwelling metallic projectiles,
* Significant valvular abnormalities,
* Pregnant women (women of childbearing potential will undergo blood or urine pregnancy testing),
* History of clinical CAD or significant epicardial coronary disease (>50% stenosis) in major coronary artery by x-ray or CT angiography unless (a) the patient underwent prior successful revascularization with percutaneous coronary angioplasty within the prior three years and (b) there are no residual lesions of >50% on the most recent coronary angiographic study.
* History of infiltrative cardiomyopathy or constrictive pericarditis,
* Cor pulmonale,
* Significant pulmonary disease,
* Estimated glomerular filtration rate (eGFR) <20ml/min,
* Any condition other than HF which could limit the ability to perform a 6MW or cardiopulmonary exercise test (CPET) test (e.g., critical peripheral vascular disease, significant orthopedic or neurological conditions),
* Any diseases other than HF which are likely to significantly alter the patient's global perception of status or quality of life over a period of 6 months.
* Significant peripheral vascular disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with and without heart failure will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mitochondrial function | Baseline
  Maximal oxidative capacity of leg muscle measured by 31P Magnetic Resonance Spectroscopy (MRS)
Skeletal muscle energetic decline during exercise | Baseline
  Creatine phosphate rate of decline (umol/g/min) during plantar flexion exercise measured by 31P MRS
Cardiac muscle energetics | Baseline
  Cardiac muscle phosphocreatine (PCr)/ adenosine triphosphate (ATP) and creatine kinase(CK) flux (umol/g/s) measured by 31P MRS

SECONDARY OUTCOMES:
Six minute walk test | Six months
  Six minute walk distance (m)
Cardiopulmonary exercise testing (CPET) | Six months
  Peak whole-body oxygen consumption rate during exercise
Clinical heart failure outcome as assessed by number of hospitalizations | Two years
Clinical heart failure outcome as assessed by time to cardiovascular death | Two years
Clinical heart failure outcome as assessed by overall mortality | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No